CLINICAL TRIAL: NCT07198282
Title: The Effect of Different Flap Closure Techniques on Postoperative Morbidity: A Randomized Controlled Trial for Impacted Third Molar Surgery
Brief Title: The Effect of Different Flap Closure Techniques on Postoperative Morbidity in Impacted Third Molar Surgery
Acronym: GMC02
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Alperen Kalyoncu, Assistant Professor, Recep Tayyip Erdogan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025/220
Record Dates: First submitted 2025-09-21; First posted 2025-09-30 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Impacted Mandibular Third Molar; Postoperative Morbidity; Oral Surgery
Keywords: Impacted third molar; Flap closure techniques; Cyanoacrylate; Sutureless technique; Surgical drain
MeSH Terms: interventions — Sutureless Surgical Procedures

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of four parallel groups to receive different flap closure techniques after impacted mandibular third molar extraction: conventional suturing, sutureless technique, surgical drain, or cyanoacrylate tissue adhesive. Each group is treated simultaneously and outcomes are compared across groups to evaluate postoperative morbidity and patient quality of life.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors evaluating postoperative morbidity (pain, swelling, trismus, wound healing) and patient quality of life (GOHAI) are blinded to the flap closure technique assigned to each participant. Surgeons and participants are not blinded due to the nature of the surgical interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Conventional Suturing (Experimental): Wound edges are approximated using 3/0 braided, non-absorbable silk sutures (Doğsan®, Turkey). Standard oral surgery closure technique.
  Interventions: Procedure: Conventional Suturing
- Sutureless Technique (Experimental): The wound is left to heal by secondary intention without any suturing material.
  Interventions: Procedure: Sutureless Technique
- Surgical Drain (Experimental): A biocompatible sterile plastic drain is placed to facilitate drainage of blood and fluids from the surgical site
  Interventions: Procedure: Surgical Drain
- Cyanoacrylate Tissue Adhesive (Experimental): Cyanoacrylate-based medical tissue adhesive (PeriAcryl®90 High Viscosity) is applied to effectively close the wound edges.
  Interventions: Procedure: Cyanoacrylate Tissue Adhesive

INTERVENTIONS:
Procedure: Conventional Suturing — Wound edges are approximated using 3/0 braided, non-absorbable silk sutures (Doğsan®, Turkey). Standard oral surgery closure technique.
  Arms: Conventional Suturing
Procedure: Sutureless Technique — The wound is left to heal by secondary intention without using any suturing material.
  Arms: Sutureless Technique
Procedure: Surgical Drain — A biocompatible sterile plastic drain is placed in the surgical site to facilitate drainage of blood and fluids, helping to reduce edema and hematoma formation.
  Arms: Surgical Drain
Procedure: Cyanoacrylate Tissue Adhesive — Cyanoacrylate-based medical tissue adhesive (PeriAcryl®90 High Viscosity) is applied to the wound edges, providing rapid polymerization and effective closure.
  Arms: Cyanoacrylate Tissue Adhesive

SUMMARY:
1. ABSTRACT This study is a randomized controlled trial comparing the clinical efficacy and safety of four different flap closure techniques in reducing postoperative morbidity (pain, swelling, trismus, wound healing) and improving patient quality of life (GOHAI) following impacted mandibular third molar extraction. The methods include conventional suturing, sutureless technique, surgical drain, and cyanoacrylate tissue adhesive, which are commonly used in oral surgery practice. The study aims to scientifically evaluate the effects of each method on patients and to determine the most appropriate clinical approach.

DETAILED DESCRIPTION:
2. INTRODUCTION Impacted mandibular third molar extraction is a commonly performed surgical procedure. Postoperative morbidity following this procedure can negatively affect patient satisfaction and quality of life. The rationale for this study is to objectively examine the role of flap closure techniques, which are an integral part of the surgical procedure, on these morbidities. The methods investigated in this research were selected due to their potential impact on wound healing and postoperative comfort.

3. PHYSICAL AND CHEMICAL CHARACTERISTICS OF THE METHODS USED

Surgical Drain Application: A biocompatible, sterile plastic tube used to drain accumulated blood and other fluids from the tissues.

Conventional Suturing Technique: Wound edges are approximated using 3/0 braided, non-absorbable silk suture (Doğsan®, Turkey). Silk suture is biologically inert and provides strong tensile strength.

Cyanoacrylate (PeriAcryl®90 High Viscosity Dental Cyanoacrylate): A cyanoacrylate-based medical tissue adhesive. Its rapid polymerization allows effective closure of wound edges.

Sutureless Technique: No material is used in this method; the wound is left to heal by secondary intention.

4. NON-CLINICAL STUDIES This study does not involve any investigational product (drug) with systemic pharmacological or toxicological effects. Therefore, no evaluation of pharmacological, toxicological, or pharmacokinetic studies in animals is relevant in this section.

5. EFFECTS ON HUMANS AND SAFETY-EFFICACY ASSESSMENT All four flap closure techniques are commonly used in oral surgery and have well-known safety profiles.

Conventional Sutures: May cause postoperative pain, swelling, and trismus. The most common adverse events are infection and bleeding.

Cyanoacrylate: Literature reports indicate it may accelerate wound healing and reduce pain. Potential adverse reactions include local irritation or allergic responses.

Surgical Drain: May contribute to wound healing by reducing edema and hematoma formation. Possible adverse events include discomfort at the incision site or infection.

Sutureless Technique: May be associated with increased postoperative pain and swelling. Wound healing may take longer compared to other methods.

This study is designed to compare the safety and efficacy of these methods using a randomized controlled methodology and to determine which method is superior in terms of patient quality of life and morbidity.

6. MARKETING EXPERIENCE The medical materials used in this study, including cyanoacrylate (PeriAcryl®90) and silk sutures (Doğsan®), are commercially available products approved by relevant regulatory authorities. None of the products have been withdrawn from the market. PeriAcryl®90 has been registered by Intertek, an MDSAP-certified auditing organization, in compliance with ISO 13485:2016 requirements.

7. SUMMARY OF DATA AND INVESTIGATOR GUIDE As the aim of this study is to compare surgical methods, it is essential that investigators understand the known benefit-risk profile of each technique. The health and safety of volunteers are the top priority.

Potential Risks and Adverse Reactions:

Expected postoperative morbidities such as pain, swelling, and trismus, as well as surgery-specific risks like infection, bleeding, and rarely nerve injury.

Precautions:

All surgical procedures will be performed according to a standardized protocol by experienced surgeons.

Volunteers will be provided with a full and understandable informed consent form detailing all risks and expectations related to the postoperative period.

Regular follow-up visits are scheduled on the 2nd and 7th days for early detection and management of potential complications.

Emergency Management:

In the event of a serious adverse event, such as life-threatening conditions or permanent disability, the protocol procedures will be immediately implemented and reported to the Turkish Medicines and Medical Devices Agency (TITCK).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-40 years.
* Patients with no systemic diseases (ASA I).
* Patients with impacted mandibular third molars indicated for extraction, with bone and/or mucosal retention, in similar positions (Pell & Gregory Class 2, Position B; Winter classification vertical or mesioangular).

Exclusion Criteria:

* Patients classified as ASA II, III, or IV.
* Known allergy to anesthetic solutions.
* Allergy to acrylate.
* Pregnant or breastfeeding women.
* Individuals with tobacco use ≥10 cigarettes/day.
* Alcohol users.
* Patients using antiplatelet agents.
* Patients using anticoagulants.
* Patients with coagulation disorders.
* Patients with immunosuppressive diseases or receiving immunosuppressive therapy.

Patients with acute pain or local infection at the surgical site.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 148 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain | 1, 3, and 7 days after surgery
  Pain intensity will be assessed using the Visual Analog Scale (VAS, 0-10 cm), where 0 = no pain and 10 = worst imaginable pain. Higher scores indicate worse outcomes.
Swelling (Edema) | 1, 3, and 7 days after surgery
  Facial swelling will be measured using standardized linear facial measurements between fixed anatomical landmarks (tragus-pogonion, tragus-oral commissure, gonion-lateral canthus). Greater values represent increased swelling.
Trismus | 1, 3, and 7 days after surgery
  Maximum interincisal mouth opening (in millimeters) will be measured using a digital caliper. Decreased values represent more severe trismus.

SECONDARY OUTCOMES:
Wound Healing | 7 and 14 days after surgery
  Wound healing will be assessed using three clinical parameters: wound edges, oral mucosa color, and wound closure, as described by Madrazo-Jiménez et al. (2016). Each parameter will be categorized as good, acceptable, or bad.
  Wound edges:
  * Good = aesthetic, clean, with well-opposed edges.
  * Acceptable = slightly irregular edges, mild bleeding or erythema.
  * Bad = irregular edges, moderate or heavy bleeding, exudate, pus, foul odor, or signs of infection.
  Oral mucosa color:
  * Good = identical to the surrounding mucosa.
  * Acceptable = similar to the surrounding mucosa.
  * Bad = erythematous.
  Wound closure:
  * Good = complete closure, no dehiscence.
  * Acceptable = 1-2 mm dehiscence.
  * Bad = dehiscence > 2 mm, open wound, keloid formation, or unaesthetic closure.
Patient Quality of Life (GOHAI) | 7 days postoperative
  Oral health-related quality of life will be assessed using the General Oral Health Assessment Index (GOHAI; score range: 12-60). Higher scores indicate better oral health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdoğan University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery, Rize, Rize Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data from this study will be made available upon reasonable request to the corresponding author after publication of the primary results. Data sharing will be for research purposes only and will require a signed data sharing agreement to ensure participant privacy and confidentiality
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Result] Kumar MS, Natta S, Shankar G, Reddy SH, Visalakshi D, Seshiah GV. Comparison between Silk Sutures and Cyanoacrylate Adhesive in Human Mucosa- A Clinical and Histological Study. J Int Oral Health. 2013 Oct;5(5):95-100. Epub 2013 Oct 26. PMID 24324311
- [Result] Sen A, Dhupar V, Akkara F. Analysing inflammatory responses after mandibular third molar extraction: a comparison of suture-less and multiple suture techniques. Oral Maxillofac Surg. 2024 Dec;28(4):1587-1594. doi: 10.1007/s10006-024-01287-2. Epub 2024 Aug 9. PMID 39117914
- [Result] Madrazo-Jimenez M, Rodriguez-Caballero A, Serrera-Figallo MA, Garrido-Serrano R, Gutierrez-Corrales A, Gutierrez-Perez JL, Torres-Lagares D. The effects of a topical gel containing chitosan, 0,2% chlorhexidine, allantoin and despanthenol on the wound healing process subsequent to impacted lower third molar extraction. Med Oral Patol Oral Cir Bucal. 2016 Nov 1;21(6):e696-e702. doi: 10.4317/medoral.21281. PMID 27475700
- [Result] Ergul S, Akar GC. Reliability and validity of the Geriatric Oral Health Assessment Index in Turkey. J Gerontol Nurs. 2008 Sep;34(9):33-9. doi: 10.3928/00989134-20080901-05. PMID 18795563
- [Result] Falci SGM, Guimaraes MTBA, Canarim NM, Falci SE, Martins OBL, de Souza GM, Galvao EL. Comparison of suture and sutureless techniques on postoperative complications after third molar surgery: a systematic review. Clin Oral Investig. 2024 Jan 25;28(1):115. doi: 10.1007/s00784-024-05518-4. PMID 38267703
- [Result] Santmarti-Oliver M, Bazal-Bonelli S, Sanchez-Labrador L, Beca-Campoy T, Perez-Gonzalez F, Cobo-Vazquez CM, Madrigal Martinez-Pereda C, Meniz-Garcia C. Cyanoacrylate versus suture as flap closure methods in mandibular third molar surgery: a split-mouth randomized controlled clinical study. Med Oral Patol Oral Cir Bucal. 2024 Jul 1;29(4):e458-e467. doi: 10.4317/medoral.26375. PMID 38907642
- [Result] Genc A, Cakarer S, Yalcin BK, Kilic BB, Isler SC, Keskin C. A comparative study of surgical drain placement and the use of kinesiologic tape to reduce postoperative morbidity after third molar surgery. Clin Oral Investig. 2019 Jan;23(1):345-350. doi: 10.1007/s00784-018-2442-x. Epub 2018 Apr 19. PMID 29675759
- [Result] Oladega AA, James O, Adeyemo WL. Cyanoacrylate tissue adhesive or silk suture for closure of surgical wound following removal of an impacted mandibular third molar: A randomized controlled study. J Craniomaxillofac Surg. 2019 Jan;47(1):93-98. doi: 10.1016/j.jcms.2018.10.018. Epub 2018 Nov 12. PMID 30501926
- [Result] Mariani P, Menditti D, Russo D, Laino L. Evaluation of the effectiveness of tube drain on postoperative discomfort in mandibular third molar surgery: prospective randomized split-mouth study. Acta Odontol Scand. 2023 Oct;81(7):528-533. doi: 10.1080/00016357.2023.2205934. Epub 2023 May 13. PMID 37177802

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-08-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT07198282/Prot_SAP_000.pdf
  • Informed Consent Form (2025-08-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT07198282/ICF_001.pdf